CLINICAL TRIAL: NCT02124239
Title: A Phase I, Multi-centre, Open-label, Uncontrolled, Non-randomised Study to Evaluate the Systemic Exposure and Safety of Ingenol Mebutate When Applied to Full Face, Balding Scalp or an Area of Approximately 250 cm2 on the Arm in Subjects With Actinic Keratosis
Brief Title: Pharmacokinetics of Ingenol Mebutate Gel in Actinic Keratosis Under Maximum Use Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0105-1034
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2016-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scalp (Experimental): Treatment of scalp with 0.027% ingenol mebutate once daily for 3 days
  Interventions: Drug: Ingenol mebutate
- Arm (Experimental): Treatment of arm with 0.06% ingenol mebutate once daily for 4 days
  Interventions: Drug: Ingenol mebutate
- Face (Experimental): Treatment of face with 0.027% ingenol mebutate once daily for 3 days
  Interventions: Drug: Ingenol mebutate

INTERVENTIONS:
Drug: Ingenol mebutate

SUMMARY:
This is an open-label, uncontrolled, non-randomised multi-centre trial in which 3 parallel groups will be enrolled. The trial includes three active treatment groups.

To be eligible for inclusion in this trial, subjects must have at least 10 clinically typical, visible, and discrete AKs on the face, balding scalp or on the arm within a contiguous area of approximately 250 cm2 of sun-damaged skin.

There will be 3 treatment groups: (1) once daily application of ingenol mebutate gel 0.027% on the full face for three consecutive days, (2) the same regimen on the balding scalp, and (3) once daily application of ingenol mebutate gel 0.06% on the arm on a treatment area of approximately 250 cm2 for four consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Following verbal and written information about the trial, the subject must provide informed consent documented by signing the Informed Consent Form prior to any trial-related procedures.2. Subjects with at least 10 clinically typical, visible and discrete AKs on the face, on approximately 250 cm2 of balding scalp or an area of approximately 250 cm2 of sun-damaged skin on the arm except the back of the hand.

3. Subject at least 18 years of age. 4. Female subjects must be of either:

* Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,

  * Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to trial treatment, to rule out pregnancy.

    5. Female subjects of childbearing potential must be willing to use effective contraception at trial entry and until completion. Effective contraception is defined as follows:
  * Oral/implant/injectable/transdermal/oestrogenic vaginal ring contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide.
  * Abstinence or partner's vasectomy are acceptable if the female agrees to implement one of the other acceptable methods of birth control if her partner changes.

Exclusion Criteria:

1. Location of the treatment area (full face, balding scalp or arm)

   * within 5 cm of an incompletely healed wound,
   * within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
2. Prior treatment with ingenol mebutate gel within the last three months.
3. Lesions in the treatment areas that have:

   * atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horns) and/or,
   * recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions).
4. Any abnormal laboratory tests that are medically significant and would impact the safety of the subjects or the interpretation of the trial results, as determined by the investigator's judgment.
5. Current enrolment or participation in an investigational clinical trial within 30 days of entry into this trial.
6. In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state).
7. Subjects with QTcF interval > 450 ms for males and 470 ms for females or other relevant pathological changes in the ECG in opinion of the investigator. These intervals apply at Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Once daily for four or five days
Peak Plasma Concentration (Cmax) | Once daily for four or five days

CONTACTS AND LOCATIONS:
Overall Officials: Alicia D Bucko, MD, Principal Investigator — Academic Dermatology Associates
Locations (1):
- Academic Dermatology Associate, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en